CLINICAL TRIAL: NCT05256485
Title: Comparing the Effect of Cognitive Behavioral Therapy, Mindfulness Based Relapse Prevention and Twelve-step Therapy in Patients With Opioid Craving
Brief Title: Comparison Between Different Psychotherapy Interventions Regarding Their Effect on Substance Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Harby (Other)
Responsible Party: Sponsor-Investigator, Sara Harby, assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPC£0521190906
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Addiction Opiate
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Standard cognitive behavioral therapy comprises approaches directed toward modifying dysfunctional thinking and behavior discussed through 8 sessions.
  mindfulness based relapse prevention is an 8-week therapy program based on:
  1. Attention to present moment experience, even if it includes craving or negative emotion.
  2. An accepting attitude towards this experience letting it be exactly as it is, without judging it or reacting to it.
  This group therapy was facilitated by an ex-addict working in El Maamora hospital.
  12-step therapy was based on strengthening conscious contact with God and awakening spirituality through prayer and meditation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cognitive behavioral therapy (Active Comparator): Standard CBT comprises an array of approaches directed toward modifying dysfunctional thinking and behavior. The two critical components are analysis of thoughts, feelings, and behaviors, as well as skills training for achieving active behavior and thought modification.
  Interventions: Behavioral: cognitive behavioral therapy,mindfulness based relapse prevention,twelve-step therapy
- mindfulness based relapse prevention (Active Comparator): MBRP training is based on a two-component process:
  1. Attention to present moment experience, even if it includes craving or negative emotion.
  2. An accepting attitude towards this experience letting it be exactly as it is, without judging it or reacting to it.
  Interventions: Behavioral: cognitive behavioral therapy,mindfulness based relapse prevention,twelve-step therapy
- twelve-step therapy (Active Comparator): 12-step therapy was based on strengthening conscious contact with God and awakening spirituality through prayer and meditation
  Interventions: Behavioral: cognitive behavioral therapy,mindfulness based relapse prevention,twelve-step therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy,mindfulness based relapse prevention,twelve-step therapy — In cognitive-behavioral therapy, participants learned that thoughts and emotions contribute to behavior, and responses to thoughts and emotions can be controlled.
  in mindfulness-based relapse prevention, participants learned to focus on the present moment experience including craving with an attitude of acceptance and non-judging.
  In twelve-step therapy, participants learned principles of acceptance, gratitude, forgiveness, tolerance, patience, humility, and honesty together with participation in different healthy ways to enrich life.

SUMMARY:
the study aim is to compare betwenn the effect of mindfulness based relapse prevention and other evidence based psychotherapy interventions regaring substance craving.

DETAILED DESCRIPTION:
In this prospective study, the population included opioid-dependent men (aged 18-50 years), some of them were admitted to El Maamora hospital and others were attendees in NA. To conduct this research, considering the drop-out rate, the list of 60 persons applying for treatment was prepared based on inclusion and exclusion criteria.

Then, three groups of 20 were randomly selected and placed in three intervention groups, group one received CBT, group two received MBRP, and group three received twelve-step therapy.

The subjects were assigned randomly to the treatment condition via a computer-generated random number with the aid of trained staff at the clinic blindly.

All participants completed the measurement scales immediately after detoxification (pre-test) and after the end of therapeutic sessions (post-test).

ELIGIBILITY:
Inclusion Criteria:

* Age: 15-50 years.
* Male gender.
* Patients meet DSM-5(3) criteria of opioid abuse.
* Had completed detoxification in a treatment center.
* Willing to give consent they will be randomly assigned to either CBT, MBRP, or twelve-step treatment group.
* Patients have dual diagnoses.
* Patients have poly-substance use disorder.

Exclusion Criteria:

* Participants with significant cognitive disorder.
* Participants with suicidal thoughts.
* Participants with any organic condition affecting stress response and so craving such as hypertension, respiratory or cardiovascular disorders.
* Participants taking any medications (e.g., antipsychotics in high doses) known to affect the stress response.
* Participants relapsed to drug abuse during therapy.

Ages: 15 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
opioid craving scale | 5 minutes
  A visual analog scale, a modification of the Cocaine Craving Scale, is a 3-item scale used to measure the opioid craving and each item is ranging from 0 to 10 (0 means no craving at all and 10 means severe craving).

SECONDARY OUTCOMES:
The Obsessive-Compulsive Drug use Scale | 15 minutes
  it measures craving in the previous ten days and includes 13 questions. Subjects should select from 5 graded options for each question based on their experiences during last week. The items were rated as follow:1) Never; 2) Rarely; 3) Sometimes; 4) Mostly and 5) Always
The desire for a drug questionnaire | 15 minutes
  it measures instant (now) craving, includes 14 questions and participants answer questions on a seven-step Likert-scale answer sheet based on what he/she feels or thinks at the moment. The items were rated as follows: 1) not at all; 2) mild; 3) mild to moderate; 4) moderate; 5) moderate to severe; 6) severe and 7) approximately complete

CONTACTS AND LOCATIONS:
Overall Officials: Tarek K Molokhia, Phd, Study Chair — professor of neuropsychiatry; Osama A Elkholy, Phd, Study Chair — professor of neuropsychiatry; Ahmed M Abdelkreem, Phd, Study Director — lecturer of neuropsychiatry; Sara A Harby, master, Principal Investigator — assistant lecturer of psychiatry
Locations (1):
- Sara Harby, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No